CLINICAL TRIAL: NCT06315673
Title: Digital Assessment of Speech and Fine Motor Control in ALS
Status: Recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: BioSensics (Industry)
Responsible Party: Principal Investigator, Andrew Geronimo, Assistant Professor, Department of Neurosurgery, Milton S. Hershey Medical Center
Other Study IDs: STUDY00024562
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Progressive Muscular Atrophy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Individuals with diagnosis of definite, probable, probable laboratory-supported, or possible ALS by revised El Escorial research criteria [2], primary lateral sclerosis (PLS), or progressive muscular atrophy (PMA).
  Interventions: Behavioral: Digital Speech and Handwriting Assessment
- Control: Individuals with no neurological or orthopedic problems that affects their speech or handwriting AND age-matched to the existing patient cohort.
  Interventions: Behavioral: Digital Speech and Handwriting Assessment

INTERVENTIONS:
Behavioral: Digital Speech and Handwriting Assessment — Subjects may complete all or some of these tests, depending on functional ability.
  * Handwriting battery
  * Pattern tracing battery
  * Speech Assessment Battery

SUMMARY:
This is a single-session, case-control study that incorporates digital tools for assessing speech and motor function in motor neuron disease. Patients with motor neuron disease (including amyotrophic lateral sclerosis (ALS), primary lateral sclerosis (PLS), and progressive muscular atrophy (PMA)) and age-matched healthy controls will be enrolled. Subjects will complete a speech and handwriting assessment during the study visit on a tablet computer (BioSensics LLC, Newton, MA). We will explore whether these digital biomarkers are sensitive to functional disease severity as reported by the ALS Functional Rating Scale - Revised (ALFRS-R) [1]. We will also compare assessment data between the patient and control groups.

DETAILED DESCRIPTION:
ALS is a progressive neuromuscular disease that causes weakness and inevitably affecting multiple motor processes within the body. To assess changes in functional mobility, clinicians and clinical investigators often rely on the ALS Functional Rating Scale - Revised (ALSFRS-R), a standardized 12-item questionnaire that has been in use for decades. Although thoroughly validated, this scale has received criticism for providing a coarse reflection of a patient's disease, scaling non-linearly within and across functional domains, and without the sensitivity to reflect day-to-day variability or small but meaningful changes.

This study includes collection of digital speech and fine motor control assessment data at a single study visit. Features extracted from this data will be compared with standard clinical disease outcome measures and also the features derived from control participant data. We will use these comparisons to explore the use of these digital assessments in capturing the range of functional changes that occur in ALS and the related motor neuron diseases of PLS and PMA that are regularly treated in the ALS clinic.

ELIGIBILITY:
Inclusion Criteria:

1. [Patient Group Only] Diagnosis of definite, probable, probable laboratory-supported, or possible ALS by revised El Escorial research criteria [Brooks2000], primary lateral sclerosis (PLS), or progressive muscular atrophy (PMA).
2. [Patient Group Only] at least minimal speech or handwriting ability

   1. ALSFRS-R speech score of 2 ("intelligible speech with repeating") or greater, OR
   2. ALSFRS-R handwriting score of 2 ("not all words are legible") or greater.
3. [Control Group Only] Possess no neurological or orthopedic problems that affects their speech or handwriting AND age-matched to the existing patient cohort.
4. 18 years of age or older;
5. Fluent in written and spoken English.

Exclusion Criteria:

1. Currently or previously enrolled in STUDY00013892 (NCT05271435)
2. Neurological or orthopedic problems (independent of their inclusionary diagnosis for the patient group) that affects their speech or handwriting
3. Pregnant or nursing woman
4. Prisoner or institutionalized individuals
5. Have any clinically relevant medical history of other disease or diseases that, in the opinion of the research team, exclude the subject from participation (including severe cognitive dysfunction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with motor neuron disease and age- and sex-matched, neurologically-healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Speaking rate during a standardized passage | baseline
  Speaking rate, in words per minute, will be determined from an audio recording of a standardized reading passage.
Residual on spiral tracing task | baseline
  Handwriting tasks include tracing of a spiral. The average residual, or deviation from the target spiral (in pixels), will be determined from the handwriting file associated with the tracing task.

SECONDARY OUTCOMES:
ALS Functional Rating Scale- Revised (ALSFRS-R) | baseline
  The ALSFRS-R measures 12 aspects of physical function, ranging from one's ability to swallow and use utensils to climbing stairs and breathing. Each function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0.
Forced vital capacity (FVC) | baseline
  FVC is collected at clinical appointments by a respiratory therapist. FVC is the volume of air that is forcefully expelled into a spirometer. FVC is expressed as a percentage (%) of predicted volume against an age, height, and ethnicity matched standard. The best result of three trials is used.
Upper motor neuron function | baseline
  Reflex testing is performed by the attending neurologist at clinical appointments. Bilateral biceps, triceps, and brachioradialis reflexes will be documented according to Modified Ashworth Scale grade 0 (no tone increase) to 4 (limb rigid). Total score for bilateral muscle groups ranges from 0 to 24.
Strength testing | baseline
  Strength testing is performed by the attending neurologist at clinical appointments. Bilateral deltoids, biceps, triceps, wrist extension, and interossei strength will be documented according to Medical Research Council (MRC) grade 0 (no power) to 5 (normal power). Total score for bilateral muscle groups ranges from 0 to 50.

CONTACTS AND LOCATIONS:
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data without identifiers may be shared with other researchers at reasonable request of the PI
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Data will become available upon publication

REFERENCES:
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847